CLINICAL TRIAL: NCT00050869
Title: Encoding a Motor Memory by Action Observation
Brief Title: Learning a Motor Task Through Observation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030074; 03-N-0074
Record Dates: First submitted 2002-12-27; First posted 2002-12-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-11-15

CONDITIONS: Healthy
Keywords: Mirror Neurons; Performance; Use-Dependent Plasticity; Attention; Premotor Cortex

SUMMARY:
Motor training results in use dependent plasticity (UDP), thought to underlie recovery of motor function after brain injury. The purpose of this protocol is to determine (a) if movement observation results in encoding of a motor memory in the primary motor cortex and (b) if observation of motor training can enhance the effects of physical training in healthy volunteers. If so, this may become an important tool in rehabilitative treatment for patients who are unable or partially able to train. We will test our hypotheses by means of focal single pulse transcranial magnetic stimulation (TMS) in a group of healthy volunteers. Our outcome measure will be the change in TMS-evoked movement direction as a function of training strategy. So far we found that this is the case in healthy volunteers (see data in analysis of the study). The purpose of this amendment is to determine if action observation can elicit the same effects in adult chronic ischemic stroke patients who have had originally significant motor weakness but recovered to the point of being able to perform the motor tasks, possibly resulting in a useful rehabilitative strategy.

DETAILED DESCRIPTION:
Motor training results in use dependent plasticity (UDP), thought to underlie recovery of motor function after brain injury. The purpose of this protocol is to determine (a) if movement observation results in encoding of a motor memory in the primary motor cortex and (b) if observation of motor training can enhance the effects of physical training in healthy volunteers. If so, this may become an important tool in rehabilitative treatment for patients who are unable or partially able to train. We will test our hypotheses by means of focal single pulse transcranial magnetic stimulation (TMS) in a group of healthy volunteers. Our outcome measure will be the change in TMS-evoked movement direction as a function of training strategy. So far we found that this is the case in healthy volunteers (see data in analysis of the study). The purpose of this protocol is to determine if action observation can elicit the same effects in adult chronic ischemic stroke patients who have had originally significant motor weakness but recovered to the point of being able to perform the motor tasks, possibly resulting in a useful rehabilitative strategy.

ELIGIBILITY:
* INCLUSION CRITERIA

Healthy volunteers and patients with thromboembolic non-hemorrhagic hemispheric lesions at least 6 months after the stroke, aged 18 to 80 years. Patients who initially had a severe motor paresis (below MRC grade 2), which subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks, and those in whom isolated thumb movements can be evoked by TMS. Handedness will be assessed by the Edinburgh inventory scale. Subjects should be able to sustain attention to the task over 30 minutes.

EXCLUSION CRITERIA

History of surgery with metallic implants or known history of metallic particles in the eye.

Patients with cardiac pacemaker, neural stimulators, cochlear implants, implanted medication pumps.

Patients with history of alcohol and drug abuse, psychiatric illness (depression, attention deficit disorder, or dementia).

Patients with severe uncontrolled medical problems (e.g. cardiovascular diseases, hypertension, diabetes mellitus, arthritis, active cancer, renal, liver, severe pulmonary diseases, infectious diseases).

Patients with epilepsy or history of loss of consciousness.

Patients with use of medications that influence synaptic plasticity as evaluated by the investigator, like antipsychotic, antidepressant acting drugs, benzodiazepines.

Patients above 80 and less than 18 years of age.

Children.

Pregnant women in the last trimester.

Patients with more than one stroke in the middle cerebral artery territory.

Patients with bilateral motor impairment.

Patients with cerebellar or brainstem lesions.

Patients unable to perform the task (wrist or elbow flexion at least MRC grade 2).

Patients with unstable cardiac arrhythmia.

Patients with h/o hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system that lower the seizure threshold or influence synaptic plasticity like neuroleptics, benzodiazepines, tricyclic antidepressants, antiepileptic medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2002-12-23; Study Completion 2007-11-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Strafella AP, Paus T. Modulation of cortical excitability during action observation: a transcranial magnetic stimulation study. Neuroreport. 2000 Jul 14;11(10):2289-92. doi: 10.1097/00001756-200007140-00044. PMID 10923687